CLINICAL TRIAL: NCT00752349
Title: To Evaluate Oral Phase Swallowing Function Using Submental Ultrasound
Status: Available | Type: Expanded Access
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeun-Chung Chang/ Department of medical imaging, National Taiwan University Hospital
Other Study IDs: 200702029R
Record Dates: First submitted 2008-09-10; First posted 2008-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Dysphagia
Keywords: Videofluoroscopic; swallowing; study; (VFSS); ultrasound
MeSH Terms: conditions — Deglutition Disorders | interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: Ultrasound — To evaluate oral phase swallowing function using submental ultrasound

SUMMARY:
Ultrasound is widely applied in many fields of medicine but less commonly used in the evaluation of tongue movement and swallowing abnormality. Fuhrman RAW reported the usefulness of using ultrasound to evaluate poor tongue coordination [1]. Peng CL stated that ultrasound could provide excellent quantitative and qualitative bases of tongue movement during swallowing using cushion-scan technique [2]. Videofluoroscopic swallowing study (VFSS) is widely accepted as the gold standard of evaluating swallowing abnormality because it is able to evaluate the whole swallowing procedure without interference of pharyngeal contraction and foreign body sensation when swallowing is examined by using a fiber-optic laryngoscope. One of the most important information that VFSS can provide is the detection of subclinical silent aspiration. The decision and management of many patients with swallowing abnormalities are usually based on the VFSS findings [3]. As shown in many reports, our experiences showed that VFSS provided extremely important information of understanding the pathophysiologic change of dysphagia due to variable etiologies, such as in patients with nasopharyngeal cancer suffering from radiation therapy [4] and in patients with stroke [5]. Using the findings of VFSS, physicians and medical staffs can make important decision whether oral feeding should be given, which safety swallowing maneuver works and what is the appropriate choices of food consistency safe to dysphagic patients. The difficulties of VFSS are usually in the transportation of paraplegic and hemiplegic patients from ward to the examining chair. The frequency and examination duration of VFSS is usually limited for avoiding unnecessary radiation exposure. Hence, ultrasound provides a role in evaluating oral condition with the benefits of convenience of transportation and availability as well as no radiation exposure. Therefore, validation of the value of ultrasound for the oral swallowing with correlation of VFSS is important to test the clinical feasibility.

Peng CL et al reported their experiences of using real-time ultrasound in the evaluation of intrinsic tongue movement [2, 6, 7]. The findings of submental ultrasound are quite different from the findings of VFSS which provides the surface information of the tongue in the swallowing of radiopaque barium sulfate bolus. Combined real-time B mode and M mode ultrasound, it was reported the potential of digital data analysis of oral phase swallowing. Kuhl V et al reported the usefulness of ultrasound in the evaluation of laryngeal elevation in patients with dysphagia [8]. They found significant decrease of laryngeal elevation in patients diagnosed as neurogenic dysphasia [8]. Casas et al successfully combined ultrasound examination and plethysmography to evaluate the swallowing condition of children with cerebral palsy [9]. The results of these studies explained the potential of ultrasound in oral swallowing and dynamic laryngeal movement.

Our experiences of VFSS showed the usefulness VFSS in diagnosing and management of patients with swallowing problem or dysphagia [4, 5, 10, 11]. To our knowledge, there was little experience of comparing between ultrasound and VFSS in patients with swallowing problem. Therefore, we conducted this study to correlate submental ultrasound and VFSS findings and tried to find out the clinical feasibility and usefulness.

Purposes: This study was to evaluate the usefulness of submental ultrasound (SM US) in oral phase swallowing in correlation with videofluoroscopic study (VFSS).

1. To compare normal volunteers and patients with swallowing abnormality with submental ultrasound.
2. To evaluate and compare patients with swallowing problem using submental ultrasound and VFSS.

Type of study: Retrospective. Time of study: Jan 2004 - July 2006.

ELIGIBILITY:
Inclusion Criteria:

* >= 20 yers

Exclusion Criteria:

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult